CLINICAL TRIAL: NCT05444439
Title: Antibiotyping and Prevalence of Virulent Genotypes Among Helicobacter Pylori and Their Impact on Response to Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nariman Zaghloul Bekhiet, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APVGHP
Record Dates: First submitted 2022-06-14; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: H Pylori Infection
Keywords: H Pylori Infection
MeSH Terms: interventions — Gastroscopy; Defecation

STUDY DESIGN:
Intervention Model Description: Histopathological examination Of gastric endoscopic biopsies Detection of cag A and vac A Genotypes by PCR in endoscopic biopsies Culture and sensitivity of endoscopic biopsies. Start empirical antibiotics regimens patient triple therapy ((levofloxacin 400 mg once , amoxicillin 1000 mg twice for 2 weeks) and (Proton pump inhibitor twice for 1 month)) then follow up by H. pylori Ag in stool.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group of naive H.Pylori infection will submitted for upper endoscopy. (Other): Upper endoscopy will be done under complete septic condition and multiple gastric biopsies from corpus and antrum will be taken for :
  1. Histopathological examination.
  2. Culture and sensitivity of endoscopic biopsies.
  3. detection of vacuolating cytotoxin A (Vac A) and cytotoxin-associated gene A (Cag A) virulent Helicobacter Pylori genotypes by polymerase chain reaction amplification(PCR).
  4. Then start empirical antibiotics regimens.
  Interventions: Genetic: detection of vacuolating cytotoxin A (Vac A) and cytotoxin-associated gene A (Cag A) virulent H.Pylori genotypes by polymerase chain reaction amplification(PCR) in gastric biopsies :; Diagnostic Test: Culture and sensitivity of endoscopic gastric biopsies:; Other: Histopathological examination endoscopic gastric biopsies:; Procedure: Upper endoscopy; Drug: empirical H.pylori regimens; Diagnostic Test: H.Pylori Ag in stool

INTERVENTIONS:
Genetic: detection of vacuolating cytotoxin A (Vac A) and cytotoxin-associated gene A (Cag A) virulent H.Pylori genotypes by polymerase chain reaction amplification(PCR) in gastric biopsies : — Extraction of DNA, using Wizard® Genomic DNA Purification Kit (Promega-USA), will be done following the manufacturer instructions. For detection of vacuolating cytotoxin A and cytotoxin-associated gene A gene, polymerase chain reaction amplification will be performed with a 9 minutes' initial denaturation at 94˚C, followed by 35 cycles of 1 minute at 94˚C, 45 seconds at 60˚C, and 45 seconds at 72˚C. Final extension will be performed for 5 minutes at 72˚C. For detection of vacuolating cytotoxin A (S1/S2, m1, m2), PCR will be performed with a 9 minutes' initial denaturation at 94˚C, followed by 35 cycles of 1 minute at 94˚C, 45 seconds at 56˚C, and 45 seconds at 72˚C. Final extension will be performed for 5 minutes at 72˚C. Amplified DNA will be analyzed by agarose gel electrophoresis. A positive sample will give bands at DNA fragment 138-bp for cytotoxin-associated gene A, at 259/286-bp for vacuolating cytotoxin A s1/s2, and 290-bp and 352-bp for m1 & m2, respectively
Diagnostic Test: Culture and sensitivity of endoscopic gastric biopsies: — During endoscopy, three biopsies will be taken from antrum and/or corpus of and will be examined by rapid urease test also known as Campylobacter-like organism test (Kimberly-Clark,USA). Culture of the bacterium on Columbia agar plus 5-7% defibrinated horse or sheep blood and selective Dent supplement under microaerophilic condition at 37degree Celsius for 3-5days.
Other: Histopathological examination endoscopic gastric biopsies: — Histological sections from the antrum and body regions will be stained with Giemsa stain. Giemsa stain working solution was prepared as follows: 40 ml Giemsa stock solution with 60 ml of distilled water. Giemsa stock solution will be prepared as follows: Giemsa powder 4 g, glycerol 250 ml and methanol 250 ml. Histological sections will be examined by a gastrointestinal pathologist to standardize the classification of gastritis. Histopathological classification will be recorded as following (acute gastritis, mild-moderate- severe chronic gastritis, Glandular atrophy or Intestinal metaplasia).
Procedure: Upper endoscopy — it will be done patient before start empirical therapy and multiple antrum and/or corpus biopsies will be taken . Patient will be fasting at least 8 hours.Upper and findings will be recorded in the report as presence of gastroesophageal reflux disease, diffuse or localised gastric and/or duodenal redness, mucosal swelling, atrophy of mucosa, nodularity, intestinal metaplasia, erosions or ulcers.
Drug: empirical H.pylori regimens — Start empirical antibiotics regimens patient triple therapy ((levofloxacin 400 mg once , amoxicillin 1000 mg twice for 2 weeks) and (Proton pump inhibitor twice for 1 month)). Follow up after 2 weeks after finishing regimen by Stool Ag in stool
Diagnostic Test: H.Pylori Ag in stool — Any symptomatic patient is above 18 years old with H pylori infection patients diagnosed by positive H pylori Ag in stool will be included.
  assessment of laboratory response, 2 weeks after finishing empirical therapy.

SUMMARY:
* Detection of primary antimicrobial susceptibility and resistance of Helicobacter Pylori infection.
* Detection of resistance and virulence genes of Helicobacter Pylori infection.
* Assessment of H pylori carcinogenicity gene.
* Evaluation of outcome and efficacy of antibiotics regimen will be used in our research.
* Evaluation of effect of other factors as diet (fatty and spicy meal), drugs as NSAIDs use, antibiotics for any cause on response of H pylori to antibiotics regimen.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection is one of the most common infections in humans, affecting more than half of the world population. New infections are thought to occur as a consequence of direct human-to-human transmission or environmental contamination.

The prevalence of the infection varies widely in rural developing areas (more than 80%) compared to urban developed ones (less than 40%), as a consequence of different socioeconomic and hygienic conditions .

The vertical mode is infection spread from ascendant to descendent within the same family, while horizontal transmission involves contact with individuals outside the family or environmental contamination.

Most individuals are infected by Helicobacter pylori during early childhood; in developing countries. Successful eradication is important to prevent the development of antibiotic resistance, as well as to reduce the number of treatments and procedures. Thus, national/ regional antibiotic resistance data could be used to guide treatment regimens for H pylori infection .

Several clinical factors associated with increased rates of antibiotic resistant H. pylori, including history of previous antibiotic exposure, increasing age, female gender, ethnicity/race, extent of alcohol use, and non-ulcer dyspepsia .

The primary antibiotic resistance of H. pylori is increasing worldwide. The overall resistance rate was found to be 4.55% for amoxicillin; 27.22% for clarithromycin; 39.66% for metronidazole; and 22.48% for levofloxacin.

Therefore, drug susceptibility result of these antibiotics is necessary to select the appropriate drug for the successful eradication of the infection.

Helicobacter pylori exhibit specific geographic distributions that are related to clinical outcomes. Despite the high infection rate of H. pylori throughout the world, the genetic epidemiology surveillance of H. pylori still needs to be improved.

ELIGIBILITY:
Inclusion Criteria:

- Any patient is above 18 years old with symptomatic H pylori infection patients diagnosed by positive H pylori Ag in stool (naïve treatment).

Exclusion Criteria:

* Patients who aren't eligible to endoscopy.
* Patients are under 18 years old
* Patient's refusal
* history of antibiotics or proton pump inhibitor use during last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
detection of pre treatment antibiotic culture and sensitivity test | up to 12 months
  During endoscopy, three biopsies will be taken from antrum and/or corpus of stomach, Biopsies will be examined for identification of H. pylori by rapid urease test also known as the Campylobacter-like organism test (Kimberly-Clark, USA). Culture of the bacterium on Columbia agar (Oxoid-UK) plus 5-7% defibrinated horse or sheep blood and selective Dent supplement (Oxoid-UK) under microaerophilic condition at 37 degree Celsius for 3-5days. So the investigators will detect prevalence and types of antibiotic H.Pylori resistance in biopsies.
detection of vacuolating cytotoxin A and cytotoxin-associated gene A virulent Helicobacter Pylori genotypes by polymerase chain reaction amplification(PCR) | up to 12 months
  Extraction of DNA, using Wizard® Genomic DNA Purification Kit (Promega-USA), will be done following the manufacturer instructions. For detection of vacuolating cytotoxin A and cytotoxin-associated gene A gene, polymerase chain reaction amplification will be performed with a 9 minutes' initial denaturation at 94˚C, followed by 35 cycles of 1 minute at 94˚C, 45 seconds at 60˚C, and 45 seconds at 72˚C. Final extension will be performed for 5 minutes at 72˚C. For detection of vacuolating cytotoxin A (S1/S2, m1, m2), PCR will be performed with a 9 minutes' initial denaturation at 94˚C, followed by 35 cycles of 1 minute at 94˚C, 45 seconds at 56˚C, and 45 seconds at 72˚C. Final extension will be performed for 5 minutes at 72˚C. Amplified DNA will be analyzed by agarose gel electrophoresis. A positive sample will give bands at DNA fragment 138-bp for cytotoxin-associated gene A, at 259/286-bp for vacuolating cytotoxin A s1/s2, and 290-bp and 352-bp for m1 & m2, respectively.
Relation of histopathological examination (gastritis classification) to clinical presentation and to resistance. | up to 12 months
  Histopathological examination of endoscopic biopsies and detect acute or chronic inflammation induced by H.pylori bacteria.

SECONDARY OUTCOMES:
Detection of diet and drugs effect on response to treatment | up to 12 months
  Detect diet intake (fatty and spicy meal), drugs use (as NSAIDs, antibiotics, proton pump inhibitors in last month) by Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Nariman Zaghloul Bekhiet, Asyut, Egypt

REFERENCES:
- [Background] Liu Y, Wang S, Yang F, Chi W, Ding L, Liu T, Zhu F, Ji D, Zhou J, Fang Y, Zhang J, Xiang P, Zhang Y, Zhao H. Antimicrobial resistance patterns and genetic elements associated with the antibiotic resistance of Helicobacter pylori strains from Shanghai. Gut Pathog. 2022 Mar 30;14(1):14. doi: 10.1186/s13099-022-00488-y. PMID 35354484
- [Background] Deng L, He XY, Tang B, Xiang Y, Yue JJ. An improved quantitative real-time polymerase chain reaction technology for Helicobacter pylori detection in stomach tissue and its application value in clinical precision testing. BMC Biotechnol. 2020 Jun 22;20(1):33. doi: 10.1186/s12896-020-00624-z. PMID 32571272
- [Background] Pokhrel N, Khanal B, Rai K, Subedi M, Bhattarai NR. Application of PCR and Microscopy to Detect Helicobacter pylori in Gastric Biopsy Specimen among Acid Peptic Disorders at Tertiary Care Centre in Eastern Nepal. Can J Infect Dis Med Microbiol. 2019 Feb 5;2019:3695307. doi: 10.1155/2019/3695307. eCollection 2019. PMID 30867850
- See also: Related Info — https://doi.org/10.3389/fcimb.2020.596371
- See also: Related Info — https://doi.org/10.1016/j.ygeno.2021.10.002